CLINICAL TRIAL: NCT04546295
Title: Effect of Smartphone Application on Reducing Localized Inflammation in Periodontal Maintenance Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0685-20-EP
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brushlink (Experimental): This group will use Brushlink and interdental cleaner. The Brushlink app downloaded to participant's cell phone. A small Brushlink device is attached to participant's toothbrush. When participant's brush their teeth, the device on the toothbrush will send information to the app on your phone about how long teeth are brushed and at what angle the toothbrush is being held against the tooth.
  Interventions: Other: Brushlink application; Other: Interproximal brush
- Water-flosser (Active Comparator): This group will brush their teeth using a waterflosser that sprays the tooth with a small jet of water.
  Interventions: Other: Water-flosser; Other: Interproximal brush
- Interproximal Brush (Placebo Comparator): This group will brush their teeth with only a toothbrush.
  Interventions: Other: Interproximal brush

INTERVENTIONS:
Other: Brushlink application — Brushlink application + Interproximal brush
  Arms: Brushlink
Other: Water-flosser — Water-flosser
  Arms: Water-flosser
Other: Interproximal brush — Interproximal brush alone

SUMMARY:
The intent of this study is to determine the effect of a smartphone application used in conjunction with interproximal cleaning on localized, inflamed periodontal pockets of periodontal maintenance patients. The hypothesis to be tested is that the use of the smartphone application will decrease clinical parameters of inflammation (probing depths, bleeding on probing) as well as the pro-inflammatory biomarker (IL-1B) as determined in gingival crevicular fluid sampling.

DETAILED DESCRIPTION:
Numerous studies have shown that high quality home care (oral hygiene) is key in achieving stability in periodontal patients. Any technology that can potentially improve a patient's home care could be instrumental in decreasing periodontal inflammation and therefore could improve a patient's overall oral health.

The clinical phase of this 6-week, randomized, single-masked, interventional clinical trial will include randomization of 66 individuals regularly attending the University of Nebraska Medical Center College of Dentistry for periodontal maintenance therapy (PMT). The inclusion criteria for the study will include patients between the ages of 40-85 years, a periodontal diagnosis of moderate-advanced chronic periodontitis, one 5-7 mm interproximal probing depth (test site) with 2 mm between inferior border of contact and gingival margin, overall good systemic health, history of regular PMT, and ownership of a smartphone device. Exclusion criteria will eliminate patients with systemic diseases that significantly affect periodontal inflammation and bone turnover, and surgical periodontal therapy within the past year. Following informed consent, patients will be randomly assigned to one of three groups (22 patients per group): one group will receive instruction in the use of an interproximal cleaner with the Brushlink® app at the test site (BL), one group will receive instruction in the use of a water-flosser at the test site, and one group will receive instruction in the use of an interproximal cleaner (IP) alone at the test site. Groups will be randomized by gender and smoking status by a clinician not involved with clinical measurements. Measurements of plaque index (PI), gingival index (GI), probing depth (PD), recession and gingival crevicular fluid (GCF) samples will obtained at baseline and 6 weeks by one of three calibrated clinicians (AK, RR, LS). During data collection, supragingival plaque will be removed (and recorded), then an absorbent paper strip will be inserted into the facial and lingual sulci of the test site for 30 seconds for collection of GCF. Following data collection, patients will be instructed to use either the interproximal brush + Brushlink®, water-flosser, or interproximal cleaner alone at the test site once daily for 6 weeks. Patients will return at 6 weeks for clinical measurements and GCF sampling. The GCF samples will be analyzed via ELISA for the inflammatory biomarker, IL-1B. Clinical data will be submitted to statistical analysis to determine differences between groups with p-values </= 0.05 being considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* a periodontal diagnosis of moderate-advanced chronic periodontitis,
* one 5-7 mm interproximal probing depth (test site) with 2 mm between inferior border of contact and gingival margin
* overall good systemic health
* history of regular PMT, and ownership of a smartphone device

Exclusion Criteria:

* systemic diseases that significantly affect periodontal inflammation and bone turnover
* surgical periodontal therapy within the past year

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 6 weeks
  Measured level of clinical attachment (periodontal ligament oncementum on the root surfaces of teeth)

SECONDARY OUTCOMES:
Bleeding on probing | 6 weeks
  Incidence of bleeding during study probing of gums.

OTHER OUTCOMES:
IL-1 levels | 6 weeks
  Pro-inflammatory biomarker (IL-1B) levels as determined in gingival crevicular fluid sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Killeen, DDS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No